CLINICAL TRIAL: NCT07237191
Title: Single Impact Versus Dual Implant Fixation of Distal Femur Extra Articular and Complete Articular Fractures in Geriatric Patients
Brief Title: Geriatric Distal Femur
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00139405
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Articular Fractures
Keywords: distal femur fractures; single implant fixation; dual implant fixation
MeSH Terms: conditions — Femoral Fractures, Distal

STUDY DESIGN:
Intervention Model Description: Adult patients with extra-articular or complete articular distal femur fractures that will be operatively treated recruited from one of the participating sites during the index hospitalization
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Implant Fixation (Other): Single implant fixation with either a precontoured lateral locking plate or an intramedullary nail which is the current standard of care.
  Interventions: Procedure: Single Implant Fixation
- Dual Implant Fixation (Other): Dual implant fixation with either a lateral locking plate plus an intramedullary nail or a lateral locking plate plus a supplemental medial plate which is the current standard of care.
  Interventions: Procedure: Dual Implant Fixation

INTERVENTIONS:
Procedure: Single Implant Fixation — Lateral precontoured 4.5 mm distal femur plate or an intramedullary nail at the surgeon's discretion. Standard-of-care techniques will be used by the surgeon for fracture reduction and implant placement.
  Arms: Single Implant Fixation
Procedure: Dual Implant Fixation — Lateral precontoured distal femur plate and either (1) an intramedullary nail or (2) a medial plate. The medial plate must span the extra-articular portion of the fracture and must have stiffness of a 3.5 mm reconstruction plate, 3.5 mm limited contact dynamic compression plate, or greater.
  Arms: Dual Implant Fixation

SUMMARY:
The goal of this clinical trial is to compare two types of surgical fixation in patients with specific kinds of distal femur fractures. The main questions it aims to answer is which operation for distal femur fractures is better for efficient return to work and everyday activities.

DETAILED DESCRIPTION:
Fractures of the distal femur are severe and common injuries sustained by older adults. Despite advances in implant technology, these injuries continue to have an unacceptably high rate of nonunion (failure to heal) of approximately 20%. This adverse outcome requires additional surgery to achieve fracture healing, which prolongs recovery and further delays return to activities of daily living and impacts quality of life. Despite numerous studies of a variety of different surgical treatment strategies, the incidence of nonunion remains high. Therefore, any novel strategy to reduce the risk of nonunion and accelerate return to activities after distal femur fracture warrants rigorous study. The goal of this study is to investigate a potential treatment for distal femur fractures that has the potential to improve the likelihood of fracture healing and accelerate return of patient function during the healing process.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 55 years
* Surgically treated displaced distal femur extra articular or complete articular fractures

Exclusion Criteria:

* Patients with injury features that preclude treatment with 2 implants
* Patients unlikely to follow-up due to homelessness, or planning follow up at another institution
* Body Mass Index (BMI) > 40
* Injury due to ground level fall
* Patient that speaks neither English or Spanish
* Patients with multisystem injuries that could preclude return to work
* < 55 years of age
* Prisoner

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of Unions | 6-week, 3, 6, 12 months
  Union, as determined by the treating surgeon, will be assessed via radiographs and documented as a dichotomous outcome (yes/no), and time to union will also be captured. Nonunion will be captured via surgeon diagnosis or return to the operating room for nonunion treatment.
Total Surgical Time - Reoperations | 6-week, 3, 6, 12 months
  The total surgical time during any reoperations will be collected from the medical record.
Number of Reoperations | 6-week, 3, 6, 12 months
  Details regarding reoperations will also be collected, whether or not the operation results in an inpatient admission.

SECONDARY OUTCOMES:
Number of Resource Utilizations | 6-week, 3, 6, 12 month
  Healthcare utilization, including all hospitalizations, emergency department visits, clinic visits, imaging, and physical therapy sessions after the index stay following injury will be documented at all follow-up visits.
Return to Work - International Physical Activity Questionnaire (IPAQ) Scores | Week 6
  Completion of the International Physical Activity Questionnaire (IPAQ). The IPAQ is a validated, self-report measure that captures detailed information about participation in a wide range of physical activities, including the number of days and amount of time spent in the previous 7 days. Responses for each type of physical activity are then transformed into the number of Metabolic Equivalent for Tasks (METs), and a METs/week is calculated for each patient. To get a continuous variable score from the IPAQ (MET minutes a week) it is considered walking to be 3.3 METS, moderate physical activity to be 4 METS and vigorous physical activity to be 8 METS. Higher scores meaning more activity.
Return to Work - International Physical Activity Questionnaire (IPAQ) Scores | Month 3
  Completion of the International Physical Activity Questionnaire (IPAQ). The IPAQ is a validated, self-report measure that captures detailed information about participation in a wide range of physical activities, including the number of days and amount of time spent in the previous 7 days. Responses for each type of physical activity are then transformed into the number of Metabolic Equivalent for Tasks (METs), and a METs/week is calculated for each patient. To get a continuous variable score from the IPAQ (MET minutes a week) it is considered walking to be 3.3 METS, moderate physical activity to be 4 METS and vigorous physical activity to be 8 METS. Higher scores meaning more activity.
Return to Work - International Physical Activity Questionnaire (IPAQ) Scores | Month 6
  Completion of the International Physical Activity Questionnaire (IPAQ). The IPAQ is a validated, self-report measure that captures detailed information about participation in a wide range of physical activities, including the number of days and amount of time spent in the previous 7 days. Responses for each type of physical activity are then transformed into the number of Metabolic Equivalent for Tasks (METs), and a METs/week is calculated for each patient. To get a continuous variable score from the IPAQ (MET minutes a week) it is considered walking to be 3.3 METS, moderate physical activity to be 4 METS and vigorous physical activity to be 8 METS. Higher scores meaning more activity.
Return to Work - International Physical Activity Questionnaire (IPAQ) Scores | Month 12
  Completion of the International Physical Activity Questionnaire (IPAQ). The IPAQ is a validated, self-report measure that captures detailed information about participation in a wide range of physical activities, including the number of days and amount of time spent in the previous 7 days. Responses for each type of physical activity are then transformed into the number of Metabolic Equivalent for Tasks (METs), and a METs/week is calculated for each patient. To get a continuous variable score from the IPAQ (MET minutes a week) it is considered walking to be 3.3 METS, moderate physical activity to be 4 METS and vigorous physical activity to be 8 METS. Higher scores meaning more activity.
Time to Walking Without an Assistive Device | 6-week, 3, 6, 12 months
  Use of an assistive device will be abstracted from the medical record and/or collected via patient interview at each follow up time point.
Prescribed Weight Bearing Status | 6-week, 3, 6, 12 months
  The prescribed weightbearing status will be captured from discharge instructions and clinic notes.
Fear of Movement -Tampa Scale for Kinesiophobia (TSK) Scores | 6-week, 3, 6, 12 months
  Tampa Scale for Kinesiophobia (TSK) will be utilized to measure fear of movement. This scale is 17 items and uses a 4-point Likert scale ranging from 'strongly disagree' to 'strongly agree'. The TSK is a validated measure for surgical and musculoskeletal patients. The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.
Health Related Quality of Life - Patient-Reported Outcomes Measurement Information System (PROMIS) Scores | 6-week, 3, 6, 12 months
  The PROMIS-29 includes seven domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities. A 5-point Likert scale is used for each question and norm-based total scores (range 0-100) have been calculated so that 50 represents the mean and one standard deviation is 10 points. Higher scores represent better function.
Global Health Status - Veterans RAND 12 Item Health Survey (VR12) Scores | 6-week, 3, 6, 12 months
  The VR-12 is a measure of global health that corresponds to seven domains: general health, physical functioning, role limitations, pain, fatigue, social functioning, and mental health. Scores range from 0 to 100. 0 indicates the lowest level of health and 100 indicates the highest level of health.
Work Productivity and Activity Impairment Questionnaire Scores | 6-week, 3, 6, 12 months
  The Work Productivity and Activity Impairment Questionnaire (WPAI) questionnaire is an instrument to measure impairments in both paid work and unpaid work. It measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Numeric Pain Rating | 6-week, 3, 6, 12 months
  Patients will be asked to rate their current pain on a visual analog scale. In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Pain Inventory (BPI) | 6-week, 3, 6, 12 months
  Pain will be assessed using the Brief Pain Inventory (BPI). The BPI is a commonly used and validated 15-item measure of pain intensity and interference with daily life. The BPI measures how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. BPI pain interference is typically scored as the mean of the seven interference items. Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain. Higher scores meaning higher pain.
Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Subscale--Pain Interference | 6-week, 3, 6, 12 months
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation - scores (range 0-100). Higher scores means a higher level of pain interference.
Presence of Post-Traumatic Arthritis (PTOA) - Kellgren Lawrence (KL) Classification | 1 year
  If PTOA is present, Kellgren Lawrence (KL) classification will be assessed by the panel of reviewers and documented. Higher scores represent worse PTOA. Grade 0 - Normal articular cartilage. Grade I - Softening and swelling. Grade II - Fragmentation and fissuring of less than 0.5 inches. Grade III - Fragmentation and fissuring of greater than 0.5 inches. Grade IV - Erosion down to the subchondral bone.
Presence of Post-Traumatic Arthritis (PTOA) - Paley Grading System (PGS) | 1 year
  If PTOA is present, the Paley Grading System (PGS) will be assessed by the panel of reviewers and documented. Higher scores represent worse PTOA. Standard joint space with no evidence of degeneration was set as Grade 0. Normal joint space with the occurrence of osteophytes, subchondral sclerosis, and cysts was set as Grade 1. Joint space narrowing was set as Grade 2. Disappeared joint space was set as Grade 3.
Geriatric Depression Scale | 6-week, 3, 6, 12 months
  This scale has been validated in many studies and is unique in that it is tailored to a geriatric population by distinguishing between undiagnosed dementia and depression. Patients will also complete this scale to measure depression as part of health-related quality of life. The Geriatric Depression Scale (GDS) includes a total score range of 0 to 15. A score of 5 or more suggests depression. A score of 6 on this scale has a 94% sensitivity and 85% specificity for Diagnostic and Statistical Manual of Mental Disorders (DSM) diagnosed depression.
Morphine Milligram Equivalents (MME) | 6-week, 3, 6, 12 months
  To evaluate pain medication as a confounder to pain scores and complications MME will be calculated at each time point. To assess MME as a confounder, MME will be compared by treatment group at each time point.
Total Surgical Time - Index Surgery | Baseline
  The total surgical time during the index surgery will be collected from the medical record
Total Hospital Days | Baseline, 6-week, 3, 6, 12 months
  Total hospital days, including the index hospitalization and any subsequent inpatient stays will be captured

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Kempton, M.D., Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No